CLINICAL TRIAL: NCT02320175
Title: Bringing I-PASS to the Bedside: A Communication Bundle to Improve Patient Safety and Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Landrigan, Professor of Pediatrics, Harvard Medical School; Research and Fellowship Director, Boston Children's Hospital Inpatient Pediatrics Service, Boston Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR-1306-03556
Record Dates: First submitted 2014-12-12; First posted 2014-12-19 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Communication
Keywords: Family Centered Rounds; Patient Safety; Errors; Adverse Events; Patient Experience; Family Engagement; Interprofessional Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention (No Intervention): Before implementation of Patient and Family Centered I-PASS.
- Post-intervention (Experimental): After implementation of Patient and Family Centered I-PASS.
  Interventions: Behavioral: Patient and Family Centered I-PASS

INTERVENTIONS:
Behavioral: Patient and Family Centered I-PASS — Patient and Family-Centered I-PASS is a bundle of communication interventions to improve the quality of information exchange between physicians, nurses, and families, and to better integrate families into all aspects of daily decision making in hospitals. The intervention included a health literacy-informed, structured communication framework for family-centered rounds; written rounds summaries for families; a training and learning program; and strategies to support teamwork and implementation.
  Arms: Post-intervention

SUMMARY:
Patient and Family-Centered I-PASS is a bundle of communication interventions to improve the quality of information exchange between physicians, nurses, and families, and to better integrate families into all aspects of daily decision making in hospitals. This project tests the hypothesis that rates of medical errors and adverse events (primary outcome), hospital experience, communication, and shared understanding will improve following implementation of Patient and Family Centered I-PASS, as compared with current practice.

DETAILED DESCRIPTION:
We conducted an intervention study on pediatric inpatient units in seven North American hospitals. Each site was assigned to one of 3 staggered waves of implementation and data collection. The Patient and Family Centered I-PASS intervention included a health literacy-informed, structured communication framework for family-centered rounds; written rounds summaries for families; a training and learning program; and strategies to support teamwork and implementation. We measured errors and adverse events (AEs) via an established systematic surveillance methodology, family experience via pre-discharge surveys, and communication processes via direct observations.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the pediatric inpatient study units of participating hospitals
* Parents/caregivers of patients less than 18 years of age who speak English, Chinese, Arabic, Russian, or Spanish
* Nurses working on these units
* Residents working on these units
* Medical students working on these units

Exclusion Criteria:

* Parents/caregivers who do not speak a study language (decided based on the 5 most commonly spoken languages across study sites; study languages include: English, Chinese, Arabic, Russian, Spanish)
* Parents/caregivers of patients greater than 18 years of age

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6478 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Landrigan, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (7):
- United States (6):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - UCSF Benioff Children's Hospital San Francisco, San Francisco, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Starmer AJ, Spector ND, Srivastava R, West DC, Rosenbluth G, Allen AD, Noble EL, Tse LL, Dalal AK, Keohane CA, Lipsitz SR, Rothschild JM, Wien MF, Yoon CS, Zigmont KR, Wilson KM, O'Toole JK, Solan LG, Aylor M, Bismilla Z, Coffey M, Mahant S, Blankenburg RL, Destino LA, Everhart JL, Patel SJ, Bale JF Jr, Spackman JB, Stevenson AT, Calaman S, Cole FS, Balmer DF, Hepps JH, Lopreiato JO, Yu CE, Sectish TC, Landrigan CP; I-PASS Study Group. Changes in medical errors after implementation of a handoff program. N Engl J Med. 2014 Nov 6;371(19):1803-12. doi: 10.1056/NEJMsa1405556. PMID 25372088
- [Background] Khan A, Coffey M, Litterer KP, Baird JD, Furtak SL, Garcia BM, Ashland MA, Calaman S, Kuzma NC, O'Toole JK, Patel A, Rosenbluth G, Destino LA, Everhart JL, Good BP, Hepps JH, Dalal AK, Lipsitz SR, Yoon CS, Zigmont KR, Srivastava R, Starmer AJ, Sectish TC, Spector ND, West DC, Landrigan CP; the Patient and Family Centered I-PASS Study Group; Allair BK, Alminde C, Alvarado-Little W, Atsatt M, Aylor ME, Bale JF Jr, Balmer D, Barton KT, Beck C, Bismilla Z, Blankenburg RL, Chandler D, Choudhary A, Christensen E, Coghlan-McDonald S, Cole FS, Corless E, Cray S, Da Silva R, Dahale D, Dreyer B, Growdon AS, Gubler L, Guiot A, Harris R, Haskell H, Kocolas I, Kruvand E, Lane MM, Langrish K, Ledford CJW, Lewis K, Lopreiato JO, Maloney CG, Mangan A, Markle P, Mendoza F, Micalizzi DA, Mittal V, Obermeyer M, O'Donnell KA, Ottolini M, Patel SJ, Pickler R, Rogers JE, Sanders LM, Sauder K, Shah SS, Sharma M, Simpkin A, Subramony A, Thompson ED Jr, Trueman L, Trujillo T, Turmelle MP, Warnick C, Welch C, White AJ, Wien MF, Winn AS, Wintch S, Wolf M, Yin HS, Yu CE. Families as Partners in Hospital Error and Adverse Event Surveillance. JAMA Pediatr. 2017 Apr 1;171(4):372-381. doi: 10.1001/jamapediatrics.2016.4812. PMID 28241211
- [Derived] Khan A, Spector ND, Baird JD, Ashland M, Starmer AJ, Rosenbluth G, Garcia BM, Litterer KP, Rogers JE, Dalal AK, Lipsitz S, Yoon CS, Zigmont KR, Guiot A, O'Toole JK, Patel A, Bismilla Z, Coffey M, Langrish K, Blankenburg RL, Destino LA, Everhart JL, Good BP, Kocolas I, Srivastava R, Calaman S, Cray S, Kuzma N, Lewis K, Thompson ED, Hepps JH, Lopreiato JO, Yu CE, Haskell H, Kruvand E, Micalizzi DA, Alvarado-Little W, Dreyer BP, Yin HS, Subramony A, Patel SJ, Sectish TC, West DC, Landrigan CP. Patient safety after implementation of a coproduced family centered communication programme: multicenter before and after intervention study. BMJ. 2018 Dec 5;363:k4764. doi: 10.1136/bmj.k4764. PMID 30518517

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-intervention | Post-intervention
Started | 3538 (Patients (n=1574); Parents (n=1222); Physicians (n=478); Nurses (n=264).) | 2940 (Patients (n=1532); Parents (n=926); Physicians (n=311); Nurses (n=171).)
Completed | 3538 (Patients (n=1574); Parents (n=1222); Physicians (n=478); Nurses (n=264).) | 2940 (Patients (n=1532); Parents (n=926); Physicians (n=311); Nurses (n=171).)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient (n=1574, n=1532) characteristics derived from hospital administrative data. Parent (n=947, n=890), Physician (n=343, n=252), Nurse (n=191, n=139) characteristics derived from self-reported survey data. Missingness (which ranged 2.0%-9.7%, except for patient race and annual household income) was similar in pre- and post-intervention cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-intervention | Post-intervention | Total
Number analyzed (Participants) | 3055 | 2813 | 5868
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: A total of 132 subjects (4.3%) were missing data on age in pre-intervention and a total of 153 subjects (5.4%) were missing data on age in post-intervention. Missing data by subject type (e.g., patient, physician) ranged from 1.2%-11.6%.
  Years
    Patient: number analyzed (Participants) | 1540 | 1492 | 3032
    Patient | 6.9 (1.7) | 7.3 (1.7) | 7.1 (1.7)
    Parent: number analyzed (Participants) | 872 | 787 | 1659
    Parent | 36.0 (1.2) | 36.3 (1.2) | 36.2 (1.2)
    Physician: number analyzed (Participants) | 334 | 249 | 583
    Physician | 28.5 (0.3) | 28.2 (0.3) | 28.4 (0.3)
    Nurse: number analyzed (Participants) | 177 | 132 | 309
    Nurse | 34.4 (0.8) | 35.5 (0.9) | 34.8 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 89 subjects (2.9%) were missing data on sex in pre-intervention and a total of 122 subjects (4.3%) were missing data on sex in post-intervention. Missing data by subject type (e.g., patient, physician) ranged from 0%-8.9%.
  Participants
    Patient: number analyzed (Participants) | 1542 | 1492 | 3034
    Patient: Female | 767 | 765 | 1532
    Patient: Male | 775 | 727 | 1502
    Parent: number analyzed (Participants) | 895 | 811 | 1706
    Parent: Female | 731 | 648 | 1379
    Parent: Male | 164 | 163 | 327
    Physician: number analyzed (Participants) | 342 | 249 | 591
    Physician: Female | 236 | 167 | 403
    Physician: Male | 106 | 82 | 188
    Nurse: number analyzed (Participants) | 187 | 139 | 326
    Nurse: Female | 171 | 124 | 295
    Nurse: Male | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Patient race derived from hospital administrative data. Parent, Physician, and Nurse race/ethnicity derived from self-reported survey data. For adult subjects, categories other than 'Hispanic or Latino' are non-Hispanic (e.g., Black = Black and Non-Hispanic). Missing data on race/ethnicity ranged from 1.6%-9.3%, except for patients (15.0% overall).
  Participants
    Patient: number analyzed (Participants) | 1360 | 1279 | 2639
    Patient: Hispanic or Latino | NA — Hospital administrative data does not provide information on ethnicity. | NA — Hospital administrative data does not provide information on ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Patient: Asian | 74 | 58 | 132
    Patient: Black | 266 | 221 | 487
    Patient: White | 708 | 600 | 1308
    Patient: Other | 312 | 400 | 712
    Parent: number analyzed (Participants) | 899 | 807 | 1706
    Parent: Hispanic or Latino | 193 | 181 | 374
    Parent: Asian | 62 | 50 | 112
    Parent: Black | 158 | 122 | 280
    Parent: White | 424 | 376 | 800
    Parent: Other | 62 | 78 | 140
    Physician: number analyzed (Participants) | 331 | 248 | 579
    Physician: Hispanic or Latino | 23 | 9 | 32
    Physician: Asian | 60 | 39 | 99
    Physician: Black | 11 | 11 | 22
    Physician: White | 226 | 176 | 402
    Physician: Other | 11 | 13 | 24
    Nurse: number analyzed (Participants) | 184 | 133 | 317
    Nurse: Hispanic or Latino | 13 | 5 | 18
    Nurse: Asian | 26 | 23 | 49
    Nurse: Black | 5 | 7 | 12
    Nurse: White | 129 | 96 | 225
    Nurse: Other | 11 | 2 | 13
Region of Enrollment [Number; unit: Participants]
  United States | 2781 | 2407 | 5188
  Canada | 274 | 406 | 680

OUTCOME MEASURES:

1. Primary Outcome: Rate of Medical Errors
Description: Our primary outcome was the rate of medical errors, including harmful errors (preventable adverse events) and non-harmful errors. Medical errors and adverse events were measured per 1000 patient-days before and after implementation of Patient and Family Centered I-PASS using an established systematic safety surveillance methodology. Trained research clinicians reviewed patient medical charts, hospital incident reports, family safety interviews, and staff reports for potential errors and adverse events. Trained physician-reviewers blinded to pre- vs. post-intervention status then categorized all suspected incidents as either adverse events, non-harmful errors, or exclusions. Adverse events that were clearly caused by a medical error were subsequently deemed preventable and all other cases were categorized as non-preventable.
Time Frame: 6 months (3 months pre, 3 months post) per site (7 sites total)
Population: Patients admitted to study units.
Measure: Number (95% Confidence Interval); unit: Medical errors per 1000 patient-days
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 1574 | 1532
Medical errors per 1000 patient-days
  Overall medical errors | 41.2 [31.2 to 54.5] | 35.8 [26.9 to 47.7]
  Non-harmful errors | 20.0 [13.2 to 30.2] | 22.0 [15.1 to 32.1]
  Harmful errors (i.e., preventable adverse events) | 20.7 [15.3 to 28.1] | 12.9 [8.9 to 18.6]

2. Secondary Outcome: Rate of Non-Preventable Adverse Events
Description: An additional measure of interest was the rate of non-preventable adverse events. Medical errors and adverse events were measured per 1000 patient-days before and after implementation of Patient and Family Centered I-PASS using an established systematic safety surveillance methodology. Trained research clinicians reviewed patient medical charts, hospital incident reports, family safety interviews, and staff reports for potential errors and adverse events. Trained physician-reviewers blinded to pre- vs. post-intervention status then categorized all suspected incidents as either adverse events, non-harmful errors, or exclusions. Adverse events that were clearly caused by a medical error were subsequently deemed preventable and all other cases were categorized as non-preventable.
Time Frame: 6 months (3 months pre, 3 months post) per site (7 sites total)
Population: Patients admitted to study units.
Measure: Number (95% Confidence Interval); unit: Non-preventable AE per 1000 patient-days
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 1574 | 1532
Non-preventable AE per 1000 patient-days | 12.6 [8.9 to 17.9] | 5.2 [3.1 to 8.8]

3. Secondary Outcome: Family Experience With Care
Description: Family experience before and after implementation. Experience was measured using a 10-15 minute survey verbally administered prior to discharge. Parents were asked to rate various aspects of their experience with care. This included experience during and after rounds, experience with written communication, experience with physicians and nurses, and overall hospital experience. The survey was developed, cognitively tested, and piloted at a non-intervention site (Boston Children's Hospital) and translated into Arabic, Chinese, Russian, and Spanish. We compared percent top-box experience ratings pre- vs. post-intervention using a GEE chi-squared test for binary outcomes, clustered by site. Top-box score was calculated as the percentage of participants that gave the top-most response for the given survey item (e.g., 5=Extremely; 5=Excellent). Missing data was accounted for through use of multiple imputations appropriate for missing data in clustered studies.
Time Frame: 6 months (3 months pre, 3 months post) per site (7 sites total)
Population: English-, Arabic-, Chinese-, Russian-, and Spanish-speaking parents/caregivers of <18-year-old patients on the study units were eligible to participate. Of these, 6-8 per week per site were randomly selected and surveyed 24 hours prior to discharge about their experiences with various aspects of communication.
Measure: Number (95% Confidence Interval); unit: Top-box percentage
Groups:
- Pre-intervention: Percent top-box score before implementation of Patient and Family Centered I-PASS.
- Post-intervention: Percent top-box score after implementation of Patient and Family Centered I-PASS.
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 651 | 573
Top-box percentage
  Understood what was said on rounds: number analyzed (Participants) | 487 | 559
  Understood what was said on rounds | 53.92 [44.60 to 62.98] | 62.84 [53.71 to 71.13]
  Explanation of changes to look out for: number analyzed (Participants) | 468 | 545
  Explanation of changes to look out for | 56.37 [47.5 to 64.85] | 58.71 [50.08 to 66.83]
  Satisfied with opportunity to ask questions on FCR: number analyzed (Participants) | 471 | 546
  Satisfied with opportunity to ask questions on FCR | 68.59 [57.73 to 77.73] | 72.11 [61.61 to 80.64]
  Medical team listened to family concerns: number analyzed (Participants) | 471 | 545
  Medical team listened to family concerns | 66.81 [56.98 to 75.36] | 71.64 [62.22 to 79.48]
  Family was included in decision making: number analyzed (Participants) | 468 | 543
  Family was included in decision making | 56.11 [46.24 to 65.52] | 58.72 [49.05 to 67.77]
  Family felt important in their role on rounds: number analyzed (Participants) | 470 | 542
  Family felt important in their role on rounds | 49.66 [41.76 to 57.57] | 56.57 [48.83 to 63.99]
  Family respectfully spoken to on rounds: number analyzed (Participants) | 469 | 544
  Family respectfully spoken to on rounds | 77.70 [70.57 to 83.51] | 78.97 [72.22 to 84.44]
  Quality of communication during morning rounds: number analyzed (Participants) | 463 | 540
  Quality of communication during morning rounds | 61.15 [51.93 to 69.62] | 66.19 [57.32 to 74.06]
  Satisfaction with frequency of updates on child: number analyzed (Participants) | 486 | 556
  Satisfaction with frequency of updates on child | 48.87 [41.17 to 56.63] | 53.83 [46.27 to 61.21]
  Quality of update explanations: number analyzed (Participants) | 484 | 554
  Quality of update explanations | 57.89 [47.53 to 67.60] | 59.64 [49.46 to 69.06]
  Inclusion in decision making later in day: number analyzed (Participants) | 478 | 553
  Inclusion in decision making later in day | 52.55 [44.49 to 60.48] | 55.05 [47.22 to 62.65]
  Frequency of written updates: number analyzed (Participants) | 484 | 559
  Frequency of written updates | 15.6 [8.90 to 25.93] | 33.7 [23.88 to 45.17]
  Understood written updates provided: number analyzed (Participants) | 206 | 404
  Understood written updates provided | 46.5 [34.17 to 59.27] | 57.86 [46.38 to 68.55]
  Usefulness of written updates: number analyzed (Participants) | 204 | 400
  Usefulness of written updates | 47.32 [36.58 to 58.3] | 49.7 [40.54 to 58.59]
  Shared understanding with doctors of medical plan: number analyzed (Participants) | 485 | 554
  Shared understanding with doctors of medical plan | 53.95 [44.56 to 63.07] | 59.16 [49.91 to 67.81]
  Doctors addressed family concerns: number analyzed (Participants) | 486 | 553
  Doctors addressed family concerns | 61.8 [52.51 to 70.3] | 65.85 [56.83 to 73.85]
  MDs made family feel important part of care team: number analyzed (Participants) | 484 | 552
  MDs made family feel important part of care team | 57.7 [45.91 to 68.67] | 60.88 [49.2 to 71.42]
  Shared understanding with nurses of medical plan: number analyzed (Participants) | 485 | 555
  Shared understanding with nurses of medical plan | 55.29 [47.98 to 62.38] | 65.41 [58.45 to 71.76]
  Nurses addressed family concerns: number analyzed (Participants) | 487 | 555
  Nurses addressed family concerns | 61.21 [53.42 to 68.46] | 70.22 [62.91 to 76.63]
  RNs made family feel important part of care team: number analyzed (Participants) | 484 | 552
  RNs made family feel important part of care team | 63.19 [53.49 to 71.93] | 70.74 [61.45 to 78.56]
  Teamwork among nurses and doctors: number analyzed (Participants) | 475 | 541
  Teamwork among nurses and doctors | 58.72 [51.90 to 65.22] | 61.43 [54.92 to 67.56]
  Understood reason for child's hospital stay: number analyzed (Participants) | 483 | 556
  Understood reason for child's hospital stay | 71.27 [60.88 to 79.82] | 71.44 [61.26 to 79.83]
  Understood requirements for child's discharge: number analyzed (Participants) | 479 | 550
  Understood requirements for child's discharge | 62.09 [53.34 to 70.13] | 65.69 [57.23 to 73.26]
  Overall quality of child's care: number analyzed (Participants) | 484 | 556
  Overall quality of child's care | 69.19 [60.27 to 76.87] | 72.79 [64.27 to 79.92]
  Quality of communication during hospital stay: number analyzed (Participants) | 482 | 557
  Quality of communication during hospital stay | 54.51 [45.85 to 62.9] | 58.7 [50.25 to 66.66]
Statistical Analysis 1: Comparison: Pre-intervention vs Post-intervention; Test type: Other — We compared percent top-box experience ratings pre- vs. post-intervention using a GEE chi-squared test for binary outcomes, clustered by site. Top-box score was calculated as the percentage of participants that gave the top-most response for the given survey item (e.g., 5=Extremely; 5=Excellent). Missing data was accounted for through use of multiple imputations appropriate for missing data in clustered studies; p < .05, GEE chi-squared test for binary outcomes

4. Secondary Outcome: Quality of Communication on Rounds
Description: Changes in quality of communication during rounds processes were assessed before and after implementation based on: (a) real-time structured direct observations of rounds (n=653) and (b) post-hoc analyses of audio-recordings of a subset of rounds observations (n=164). Research assistants conducted 1-hour weekly in-person rounds observation sessions per site, simultaneously completing a real-time assessment tool for each patient and audio-recording rounds. Site research clinicians blinded to pre- vs. post-intervention status conducted post-hoc analyses of a subset of rounds audio recordings using a structured assessment tool to measure rounding team adherence. Percent top-box ratings pre- vs. post-intervention were compared using a GEE chi-squared test for binary outcomes, clustered by site. Top-box score was calculated as the percentage of participants that gave the top-most response (e.g., 5=Excellent). Missing data were accounted for through use of multiple imputations.
Time Frame: 6 months (3 months pre, 3 months post) per site (7 sites total)
Population: Observations and audio-recordings of rounds were conducted at each site for one hour at a time on a randomly selected day each week. A median of 3 (IQR 2,5) patients were observed and recorded per session. Of these, 2 patients per week per site were randomly selected for post-hoc analysis.
Measure: Number (95% Confidence Interval); unit: Top-box percentage
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 305 | 348
Top-box percentage
  Family-centered rounds occurred for this patient | 72.2 [53.5 to 85.4] | 82.8 [64.9 to 92.6]
  Nurse engagement | 20.4 [7.04 to 46.6] | 35.5 [17.0 to 59.6]
  Family engagement | 55.6 [32.9 to 76.2] | 66.7 [43.0 to 84.1]
  Written summary provided to family | 17.8 [4.7 to 48.6] | 53.6 [27.4 to 78.0]
  Family expressed concerns at start of rounds: number analyzed (Participants) | 81 | 81
  Family expressed concerns at start of rounds | 18.2 [5.7 to 45.3] | 37.7 [17.6 to 63.3]
  Family reporting of illness severity: number analyzed (Participants) | 81 | 83
  Family reporting of illness severity | 28.8 [13.1 to 52.1] | 43.5 [23.8 to 65.4]
  Family synthesis (i.e., reading back) of key items: number analyzed (Participants) | 79 | 83
  Family synthesis (i.e., reading back) of key items | 4.7 [0.7 to 25.2] | 26.5 [26.5 to 12.7]
  Effective use of plain language by providers: number analyzed (Participants) | 81 | 83
  Effective use of plain language by providers | 28.8 [9.2 to 61.5] | 34.7 [12.6 to 66.3]

5. Secondary Outcome: Shared Understanding Between Parent, Resident, and Nurse
Description: Shared understanding between parent, resident, and nurse was measured before and after implementation of the Patient and Family Centered I-PASS intervention.
Time Frame: 6 months (3 months pre, 3 months post) per site (7 sites total)
Population: These data were collected but final analyses are still pending. The shared understanding measure was a novel secondary measure in this study, and the analysis was more complex than initially anticipated. Therefore, the number of participants analyzed is currently 0.
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time on study unit, from admission to discharge, on average approximately 5 days.
Description: Please see 'Rate of Medical Errors' and 'Rate of Non-Preventable Adverse Events' for detailed results on rates of adverse events pre- and post-intervention.
Arm/Group | Pre-intervention | Post-intervention
All-Cause Mortality (participants affected / at risk) | 0/1574 | 0/1532
Serious Adverse Events (participants affected / at risk) | 165/1574 | 95/1532
Other Adverse Events (participants affected / at risk) | 0/1574 | 0/1532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-intervention (N=1574) | Post-intervention (N=1532)
Serious Adverse Events (General disorders) | 165 (192) | 95 (112) — These adverse events are not related to the intervention and are adverse events captured system-wide as part of the study's main outcome.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-intervention (N=1574) | Post-intervention (N=1532)
Other Adverse Events (General disorders) | 0 (0) | 0 (0) — These adverse events are not related to the intervention and are adverse events captured system-wide as part of the study's main outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes